CLINICAL TRIAL: NCT03751748
Title: Flow Regulation by Opening the Septum in Patients With Heart Failure (FROST-HF) Trial
Brief Title: Flow Regulation by Opening the Septum in Patients With Heart Failure Trial
Acronym: FROST-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Sinai Health System (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC201809
Record Dates: First submitted 2018-11-14; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure With Normal Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, sham controlled, single blind with objective end points.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Sham Comparator): Sham procedure to include cardiac catheterization and hemodynamic. Ongoing management at the discretion of the treating physician. Patient to undergo
  Interventions: Device: Sham procedure
- AFR arm (Experimental): Implantation of Occlutech atrial flow regulator (AFR) device
  Interventions: Device: AFR implantation

INTERVENTIONS:
Device: AFR implantation — Implantation of atrial flow regulator (AFR) device
  Arms: AFR arm
Device: Sham procedure — Sham procedure to include cardiac catheterization and hemodynamic. Ongoing management at the discretion of the treating physician. Patient to undergo
  Arms: Control arm

SUMMARY:
To investigate the safety and efficacy of a novel atrial flow regulator (AFR) device in patients with heart failure and preserved ejection fraction.

DETAILED DESCRIPTION:
The study will allow us to demonstrate the safety of the AFR device as well as determine the clinical response of the therapeutic intervention. In addition, the invasive exercise hemodynamics will provide objective data for the changes in the cardiac hemodynamics and delineate underlying mechanisms of creating a permanent inter atrial shunting.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age > 40 years
* LVEF > 45% documented within the last 3 months.
* NYHA class ≥II status or 6MWT distance <80% predicted.
* Left atrial enlargement
* PCWP ≥25 mmHg during supine bicycle exercise on hemodynamic monitoring.
* Left atrial pressure greater than right atrial pressure by ≥5 mmHg on hemodynamic monitoring.

Exclusion Criteria:

* Recent MI, PCI or CABG
* Untreated CAD with indication for revascularization
* Recent stroke, pulmonary embolism or major surgery
* Uncontrolled atrial fibrillation
* H/O cardiomyopathy (hypertrophic, restrictive, infiltrative) or pericardial disease
* Inability to perform a 6-minute walk test.
* Clinically significant valvular disease
* Uunsuitable for study participation at investigator discretion.
* Severe COPD, Anemia or morbid obesity
* Uncontrolled hypertension
* Women of child bearing age
* RA pressure >15 mmHg or PVR >4 wood units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
6MWT | 12 months
  Six minute walk test at 12 months

SECONDARY OUTCOMES:
MACE | 12 months
  Composite of cardiac death, heart failure hospitalization and worsening heart failure
Cardiac death | 12 months
  Death from a cardiac cause (myocardial infarction, sudden death)
Congestive heart failure (CHF) | 12 months
  Heart failure hospitalization, worsening heart failure
Quality of Life (QOL) | 12 months
  QOL as per KCCQE questionaire

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - St. Michael's hospital, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No